CLINICAL TRIAL: NCT00373464
Title: Etoricoxib for Routine Post-operative Pain Prophylaxis in Laparoscopic Gynaecologic Surgery With Expected Need of Post-operative Opioids
Brief Title: Etoricoxib for Routine Post-operative Pain Prophylaxis in Laparoscopic Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ullevaal University Hospital (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry); University of Oslo (Other)
Organization: Oslo University Hospital (Other)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 2005-003078-92
Record Dates: First submitted 2006-09-06; First posted 2006-09-08 (Estimated); Last update posted 2011-07-01 (Estimated); Status verified 2005-08

CONDITIONS: Hysterectomy; Tubal Excision; Ovariectomy; Postoperative Pain
Keywords: Postoperative pain; Opioid; Etoricoxib; Ketorolac; Laparoscopic Surgery; Surgical Procedures, Gynecologic
MeSH Terms: conditions — Pain, Postoperative | interventions — Etoricoxib

INTERVENTIONS:
Drug: etoricoxib

SUMMARY:
The aim of this trial is to compare if a single dose of oral etoricoxib 120 mg will have equal post-operative analgesic efficacy as an optimal regiment of intravenous ketorolac 30 mg + 30 mg during the first 18 hours (+/- 1 hour) after gynaecologic laparoscopic surgical procedures, where the need for post-operative opioid is expected.

DETAILED DESCRIPTION:
Postoperative pain can contribute to reduce the patient well-being and, if it is pronounced, delay rehabilitation and increase the total cost for nursing and treatment.

As quite extensive surgical procedures presently are being undertaken on an ambulatory basis the need for adequate post-operative pain prophylaxis is stressed. Pain and nausea/vomiting are the most frequent causes of delayed discharge or unanticipated admission to hospital stay after ambulatory surgery (1). As opioids for postoperative pain relief have a lot of unwanted side-effects (e.g. nausea, vomiting, sleepiness, obstipation, disturbed physiological sleep [2]), it has been shown beneficial, both in terms of cost-effectiveness and patient satisfaction, to reduce the need of opioids in post-operative setting by other means (i.e. non-opioid) methods of pain-relief. The concept of multimodal, non-opioid pain prophylaxis and treatment is being advocated as optimal after ambulatory surgery. The most important modes of non-opioid pain prophylaxis, at present, is paracetamol, non-steroidal anti-inflammatory drugs (NSAIDs) and local anaesthesia. The best result is achieved when these different modes are used together in a prophylactic manner; the need of rescue opioid analgesics may be reduced by 20-50% and in many cases diminish (3). It has been shown in many studies that the NSAID is an important component in routine post-operative pain prophylaxis, e.g. NSAID in combination with paracetamol provides better analgesic effect than paracetamol alone, and may be equianalgesic to a small-medium dose of opioid (2).

There are four problems with NSAIDs when used for routine pain prophylaxis in ambulatory surgery/anaesthesia: increased bleeding tendency, gastrointestinal ulceration, renal failure and anaphylactic reactions (2-4).

There are definite potential benefits with etoricoxib in ambulatory setting (5-7): Due to cox-II selectivity there is no concern of increased bleeding tendency; thus the drug can be given pre-operatively. It is a potent, oral coxib; thus cheaper and more simple than IV NSAIDs. It has a long duration of effect; thus the need of patient attention is reduced because the first dose lasts for 24 h and a single daily dose will be optimal further on.

It has a lower potential of gastrointestinal ulceration, thus may be used in some patients where conventional NSAIDs may be contraindicated.

It has so far not been shown to have harmful cardiovascular effects in prospective studies of continuous use for at least 12 months in patients with increased risk of cardiovascular complications (ref 8: Edge study).

Study rationale: Etoricoxib has so far been compared with traditional oral NSAIDs and oral coxibs for postoperative pain prophylaxis. However, in many clinical situations the use of pre-operative conventional NSAIDs is not recommended due to the risk of preoperative bleeding. These patients are usually given IV ketorolac during the last part of the procedure as the most efficient alternative for post-operative pain prophylaxis.

It will be of great interest to compare this practice with the use of oral etoricoxib given pre-operatively. If the analgesic quality of an adequate dose etoricoxib is comparable to a ketorolac regimen, the etoricoxib approach will have a lot of potential benefits: simple, cheap, earlier start of analgesia, more longlasting analgesia and less risk of postoperative bleeding and gastrointestinal ulcer. If successful, a single pre-operative dose of etoricoxib may be a routine measure in a majority of all ambulatory surgery patients.

Hypotheses: A single dose pre-operative of oral etoricoxib 120 mg will have equal post-operative analgesic efficacy as an optimal regimen of IV ketorolac 30 mg + 30 mg during the first 18 h( +/- 1 h) after gynaecologic laparoscopic surgical procedure, where the need for post-operative opioid is expected.

Bibliography:

1. Chung F, Mezei G: Adverse outcomes in ambulatory anesthesia. Can. J Anaesth. 1999; 46:R18-R34.
2. Dahl V, Raeder JC: Non-opioid postoperative analgesia. Acta Anaesthesiol. Scand. 2000; 44:1191-203.
3. Dahl V, Raeder JC, Drosdal S, Wathne O, Brynildsrud J: Prophylactic oral ibuprofen or ibuprofen-codeine versus placebo for postoperative pain after primary hip arthroplasty. Acta Anaesthesiol. Scand. 1995; 39:323-6.
4. Rawal N: Postoperative pain management in day surgery. Anaesthesia 1998; 53 Suppl. 2: 50-2.
5. Chang DJ, Desjardins PJ et al. The analgesic efficacy of etoricoxib compared with oxycodone/acetaminophen in an acute post-operative pain model. Anest. Analg. 2004; 99; 807-15.
6. Cochrane DJ, Jarvis B et al. Etoricoxib. Drugs 2003; 62:2637-51.
7. Malmstrøm K, Sapre A et al. Etoricoxib in acute pain associated with dental surgery. Clin. Ther. 2004; 26:667-79.
8. The EDGE study: MSD preliminary communication.

ELIGIBILITY:
Inclusion Criteria:

* Patients (American Society of Anaesthesiologists [ASA] I and II) due for elective, laparoscopic gynaecologic surgery with the expected need for post-operative opioids: hysterectomy, removal of tube(s) and/or ovarium.
* Written informed consent.
* Weight between 50 and 120 kg.

Exclusion Criteria:

* Patients who use nonsteroidal anti-inflammatory agents (NSAIDs) in the last 48 hours (h) before surgery or are allergic to NSAIDs. Patients using steroids, anti-emetic drugs, or opioids in the last 48 h before surgery.
* Sensitivity to the study drug or its components.
* Cardiovascular risk conditions: heart failure, unstable hypertension, coronary artery disease (i.e. angina, previous myocardial infarction, previous coronary artery bypass surgery).
* Cerebrovascular disease.
* Other applicable exclusion criteria.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126
Dates: Start 2006-03; Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Equal opioid consumption in both groups postoperatively

SECONDARY OUTCOMES:
Equal visual analogue scale (VAS) and verbal rating scale (VRS) in the first 4 hours

CONTACTS AND LOCATIONS:
Overall Officials: Johan Ræder, Prof.MD,PhD, Study Director — Ullevaal University Hospital; Harald Lenz, MD, Principal Investigator — Ullevaal University Hospital
Locations (1):
- Ullevaal University Hospital, Oslo, Oslo County, Norway